CLINICAL TRIAL: NCT05520463
Title: A Prospective Randomized Comparison of Fluoroscopy and Ultrasound Guidance for Sacral Lateral Branch Radiofrequency Ablation
Brief Title: Fluoroscopy Versus Ultrasound Guidance for Sacral Lateral Branch Radiofrequency Ablation
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Diskapi Teaching and Research Hospital (Other)
Responsible Party: Principal Investigator, Halil Cihan Kose, Principle Investigator, Diskapi Teaching and Research Hospital
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: 127/23
Record Dates: First submitted 2022-08-24; First posted 2022-08-30 (Actual); Last update posted 2023-07-07 (Actual); Status verified 2023-07

CONDITIONS: Sacroiliac Joint Arthritis; Back Pain
MeSH Terms: conditions — Sacroiliitis; Back Pain

STUDY DESIGN:
Who Masked: Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Ultrasound guided sacral lateral branch radiofrequency ablation (Experimental): Patients in this group will receive sacral lateral branch radiofrequency ablation under ultrasound guidance.
  Interventions: Procedure: Sacral lateral branch radiofrequency ablation under ultrasound guidance
- Fluoroscopy guided sacral lateral branch radiofrequency ablation (Active Comparator): Patients in this group will receive sacral lateral branch radiofrequency ablation under fluoroscopy guidance.
  Interventions: Procedure: Sacral lateral branch radiofrequency ablation under fluoroscopy guidance

INTERVENTIONS:
Procedure: Sacral lateral branch radiofrequency ablation under ultrasound guidance — Sacral lateral branch radiofrequency ablation will be performed under ultrasound guided approach.
  Arms: Ultrasound guided sacral lateral branch radiofrequency ablation
Procedure: Sacral lateral branch radiofrequency ablation under fluoroscopy guidance — Sacral lateral branch radiofrequency ablation will be performed under fluoroscopy guided approach.
  Arms: Fluoroscopy guided sacral lateral branch radiofrequency ablation

SUMMARY:
Sacroiliac joint is a diarthroidal and synovial joint that receives sensory innervatin by the sacral lateral branches ( commonly S1-3, with variable contributions from L5 dorsal ramus and S4 lateral branch). Sacral lateral branch radiofrequency ablation and block techniques are widely used for the management of sacroiliac joint pain. With the increasing use of ultrasound technology in pain medicine, the ultrasound guided approaches gained popularity. To our knowledge, there are no randomized controlled trials comparing the ultrasound and fluoroscopy approaches for sacral lateral branch radiofrequency ablation. This study aims to compare the ultrasound and fluoroscopy guidance techniques for sacral lateral branch radiofrequency ablation.

ELIGIBILITY:
Inclusion Criteria:

* Low back pain due to sacroiliac joint dysfunction >6 months with a score ≥ 4 on a numeric rating scale.

  * 50% pain relief after prognostic sacral lateral branch block
* At least 3 positive physical examination maneuvers [ Faber ( flexioni abduction and external rotation), POSH (posteripr shear), REAB ( resisted abduction), Gaenslen's test, Distraction test]
* Refractory to conservative therapy

Exclusion Criteria: The exclusion criteria were;

* Uncontrolled psychiatric or neurological illness
* Sacroiliac joint pain due to other disorders,
* Lumbar radiculopathy
* Rheumatological diseases
* Systemic active infections
* Malignancies, previous surgery on the affected sacroiliac joint,
* History of traumatic hip injury,
* History of bleeding disorders,
* Platelet values < 150.000 / µl,
* Sacroiliac joint injection within the preceding 3 months,
* Allergy to local anesthetics and steroids,
* Pregnancy, inability to concent, Implanted pacemaker or defibrilator.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 60 (Actual)
Dates: Start 2022-09-01 (Actual); Primary Completion 2023-06-25 (Actual); Study Completion 2023-07-05 (Actual)

PRIMARY OUTCOMES:
Change in pain numerical rating score from baseline | 3 months
  The numerical rating score (NRS) will be used to assess the severity of pain felt by a patient. . The patient rates pain on a scale of 0 to 10; 0 represents 'no pain' and 10 ,represents 'worst pain imaginable'

SECONDARY OUTCOMES:
Performance time | During the procedure
  Radiofrequency ablation performance time will be recorded from the time the first image is obtained, until the procedure is completed
Patient satisfaction | At 3 months
  Changes in overall satisfaction will be assessed using a 5-point Likert scale. (1, very dissatisfied; 2, dissatisfied; 3, neutral; 4, satisfied; 5, very satisfied).
Pain medication use | At 3 months
  Mean change in analgesic consumption is assessed using QAQ, a tool designed to record patient-reported pain medication use. The higher score indicates higher pain medication use
Success rate | At 3 months
  Proportions of reporting >50% pain relief.
Functional disability | At 1 and 3 months
  Change in Oswestry Disabilit Index ( Scale 0-100). 0 point is equated with no disability and 100 point is maximum disability possible
Quality of life ( SF-36) | At 1 and 3 months
  Quality of life (QoL) will assessed via SF-36, which consists of 36 items ad 2 summary values for Physical Component Summary ( PSC) and Mental Component Summary (MSC). Subscale scores range from 0 to 100, with 100 being the most positive QoL in that area and 0 the lowest;
The number of needle passess | During the procedure
  The number of attempts during the performance will be analysed.

CONTACTS AND LOCATIONS:
Locations (1):
- Health Science University Diskapi Yildirim Beyazıt Training and Research Hospital, Yenimahalle, Ankara, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: No
Findings of this study will be available from the principle investigator upon reasonable request.

REFERENCES:
- [Background] Finlayson RJ, Etheridge JB, Elgueta MF, Thonnagith A, De Villiers F, Nelems B, Tran DQ. A Randomized Comparison Between Ultrasound- and Fluoroscopy-Guided Sacral Lateral Branch Blocks. Reg Anesth Pain Med. 2017 May/Jun;42(3):400-406. doi: 10.1097/AAP.0000000000000569. PMID 28178092
- [Background] Cox RC, Fortin JD. The anatomy of the lateral branches of the sacral dorsal rami: implications for radiofrequency ablation. Pain Physician. 2014 Sep-Oct;17(5):459-64. PMID 25247902